CLINICAL TRIAL: NCT04750785
Title: Choroideremia Health Outcomes
Brief Title: A Study to Assess Choroideremia (CHM) Health Outcomes
Status: Completed | Type: Observational
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Other Study IDs: US-CHM-11722
Record Dates: First submitted 2021-02-08; First posted 2021-02-11 (Actual); Last update posted 2021-10-14 (Actual); Status verified 2021-10

CONDITIONS: Choroideremia
MeSH Terms: conditions — Choroideremia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- All Participants: Participants who have been diagnosed with CHM will be enrolled.
  Interventions: Other: No Intervention

INTERVENTIONS:
Other: No Intervention — Administered as specified in the treatment arm.

SUMMARY:
The primary objectives of this study are to describe disease progression and severity by age in participants with CHM, to assess health-related quality-of-life, resource utilization and work productivity, and to assess quality-of-life, work productivity, and impact on daily activities in caregivers of participants with CHM at different stages of disease progression.

ELIGIBILITY:
Key Inclusion Criteria:

Physician Participants

1. At least 60% of time spent in direct participant care.
2. Board-certified or eligible with a Specialty in Ophthalmology, such as Retinal Specialist, IRD Specialist, Retinal Surgeon.

Patient Participants

1. CHM diagnosis confirmed via genetic testing.
2. Include any minimal disease severity requirement.
3. Participant has at least one record of visual acuity measurement in the past 24 months, OR has be assigned by the treating clinician as having severe VA impairment of blind/legally blind by using one of the following methods: finger counting, hand movement, light perception / no light perception.

Key Exclusion Criteria:

Physician Participants

a. Participating physicians must not be affiliated with an approved management organization.

Patient Participants

a. Participants who received gene therapy or any other investigational treatment and participants who do not agree to informed consent.

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply.

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Study Population: Participants who have been diagnosed with CHM. A minimum of approximately 50% of the participants will have an associated caregiver who will participate.
  Participating physicians will enroll participants for inclusion in the study.
Sampling Method: Non-Probability Sample
Enrollment: 46 (Actual)
Dates: Start 2020-12-15 (Actual); Primary Completion 2021-09-27 (Actual); Study Completion 2021-09-27 (Actual)

PRIMARY OUTCOMES:
Time to Disease Progression by Age in Participants with CHM | Up to 8 months
Best Corrected Visual Acuity by Age | Up to 8 months
  Best corrected visual acuity will be used as an indicator to assess disease severity.
Participants with CHM: EuroQol- 5 Dimension- 5 Level (EQ-5D-5L) Score | Up to 8 months
  EQ-5D is a self-report measure of health for clinical and economic appraisal. Participants complete the 5-level (no problems, slight problems, moderate problems, severe problems, and extreme problems), 5-dimension (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression) questionnaire concerning their current health state. A unique EQ-5D-5L health state scale ranges from 0 to 100 and is defined by combining 1 level from each of the 5 dimensions. Participants indicate their current health status by marking on a continuum ranging from 100 (best imaginable health state) to 0 (worst imaginable health state). The questionnaire will be implemented only one time per person in the study duration.
Participants with CHM: Health Utilities Index (HUI3) Score | Up to 8 months
  Health Utilities Index (HUI3) is a family of generic preference-based systems for measuring comprehensive health status and health-related quality of life (HRQL). HUI® provides descriptive evidence on multiple dimensions of health status, a score for each dimension of health, and a HRQL score for overall health. Health dimensions include vision, hearing, speech, ambulation/mobility, pain, dexterity, self-care, emotion and cognition. Each dimension has 3- 6 levels. HUI® systems describe almost a million unique health states. HUI3 score ranges from 0.36 (worst) to 1 (best). The questionnaire will be implemented only one time per person in the study duration.
Participants with CHM: Work Productivity and Activity Impairment (WPAI) Score | Up to 8 months
  The Work Productivity and Activity Impairment (WPAI) is a 6 questionnaire scale used to measure lost work productivity and impairment in daily activities over the past seven days. The WPAI yields four types of scores: 1. Absenteeism 2. Presenteesism 3. Work productivity loss 4. Activity Impairment, ranging from 0-100%. Higher numbers indicate greater impairment and less productivity. The questionnaire will be implemented only one time per person in the study duration.
Participants with CHM: Visual Function Questionnaire (VFQ-25) Score | Within 8 months
  VFQ-25 is a reliable and valid 25-item version of the 51-item National Eye Institute Visual Function Questionnaire (NEI-VFQ). It is especially useful in settings such as clinical trials, where interview length is a critical consideration. The global score derives from the summary of the scores deriving from each question. The total score has a minimum value "0" considered as the worst visual functionality, and the maximum value "100" considered as the better visual functionality. The questionnaire will be implemented only one time per person in the study duration.
Resource Utilization in Participants with CHM | Up to 8 months
  Healthcare Resource Utilization will be assessed by number of primary care provider visits, specialist visits, urgent care visits, emergency room (ER) visits, hospitalizations, and rehabilitation visits in past 12 months when stratified by all-cause & CHM-related.
Caregivers of Participants With CHM: Caregiver-reported Depression Via Patient Health Questionnaire-9 (PHQ-9) Score | Up to 8 months
  PHQ-9 can be used to screen for or diagnose depression, as well as measure depression severity. The PHQ-9 measures frequency of depression symptoms, with items scored on a 4-point scale (not at all=0 to nearly every day=3). The total score ranges from 0-27 where 0 is no depression and 27 is severe depression. The questionnaire will be implemented only one time per person in the study duration.
Caregivers of Participants With CHM: Caregiver-reported Anxiety Via General Anxiety Disorder-7 (GAD-7) Score | Up to 8 months
  GAD-7 is a 7-item questionnaire that is used for screening, diagnosing, monitoring, and measuring the severity of anxiety. Each item can be answered on a 4 point scale running from 0= 'not at all sure' to 3= 'nearly every day'. The total score ranges from 0-21 where 0 is no anxiety and 27 is severe anxiety. The questionnaire will be implemented only one time per person in the study duration.
Caregivers of Participants With CHM: Caregiver Reaction Assessment (CRA) Score | Up to 8 months
  Caregiver Reaction Assessment is a 24-item instrument assessing positive and negative aspects of caregiving (esteem, lack of family support, finances, schedule, and health). Each item is rated on a 1 to 4 scale. 1 (not at all) 2 (somewhat) 3 (quite a bit) 4 (completely). The questionnaire will be implemented only one time per person in the study duration.
Caregivers of Participants With CHM: Work Productivity and Activity Impairment Caregiver (WPAI-CG) Score | Up to 8 months
  WPAI-CG is a 6 questionnaire scale used to measure lost work productivity and impairment in daily activities over the past seven days. The WPAI yields four types of scores: 1. Absenteeism 2. Presenteesism 3. Work productivity loss 4. Activity Impairment, ranging from 0-100%. Higher numbers indicate greater impairment and less productivity. The questionnaire will be implemented only one time per person in the study duration.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (8):
- United States (8):
  - Research Site, Los Angeles, California
  - Research Site, San Francisco, California
  - Research Site, Coral Gables, Florida
  - Research Site, Gainesville, Florida
  - Research Site, Portland, Oregon
  - Research Site, Pittsburgh, Pennsylvania
  - Research Site, Dallas, Texas
  - Research Site, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
In accordance with Biogen's Clinical Trial Transparency and Data Sharing Policy on http://clinicalresearch.biogen.com/
URL: https://vivli.org/